CLINICAL TRIAL: NCT04684537
Title: Effect of Ultrasound-guided Piriformis Muscle Corticosteroid Injection Versus Extracorporeal Shock Wave Therapy for Piriformis Syndrome
Brief Title: Effect of Ultrasound-guided Piriformis Muscle Corticosteroid Injection Versus Extracorporeal Shock Wave Therapy for Piriformis Syndrome: a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200715R; 2021SKHADR033 (Other Grant/Funding Number: Shin Kong Wu Ho-Su Memorial Hospital)
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Piriformis Syndrome; Corticosteroid Injection; Extracorporeal Shockwave Therapy; Therapeutic Exercise
Keywords: Piriformis syndrome; ultrasound-guided intervention; corticosteroid injection; extracorporeal shockwave therapy; therapeutic exercise
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave group (Active Comparator): each subject will receive extracorporeal shockwave therapy
  Interventions: Procedure: Extracorporeal shockwave therapy (ESWT)
- Injection group (Active Comparator): each subject will receive ultrasound-guided piriformis corticosteroid injection
  Interventions: Procedure: Ultrasound-guided piriformis steroid injection

INTERVENTIONS:
Procedure: Extracorporeal shockwave therapy (ESWT) — The therapy will be performed with the focused piezoelectric shockwave (F10G4 Richard Wolf GmbH, Germany). The patient will be kept in the hip flexion, adduction and internal rotation position. After sonography-guided localization of the affected muscle and identification of the trigger point by the participant, ultrasound gel is applied to the skin and the applicator couple is placed with an impulse energy flux density of 0.456-0.882 mJ/mm2 for 3500 impulses.
  Arms: Shockwave group
Procedure: Ultrasound-guided piriformis steroid injection — all the participants will receive ultrasound-guided piriformis injection with 10 mg triamcinolone and 1 c.c. 1% lidocaine for one time.
  Arms: Injection group

SUMMARY:
In this study, the investigators aim to compare the effect of extracorporeal shockwave therapy with ultrasound-guided piriformis coticosteroid injection in treatment of PS.

DETAILED DESCRIPTION:
Piriformis syndrome (PS) is one of the common etiology of low back pain. The cause of PS is due to myofascial syndrome of piriformis muscle, leading to piriformis muscle spasm, string-like taut band, and trigger point. Consequently, it may compresses the sciatic nerve which arise from sciatic notch and passes under the piriformis muscle. Conservative treatment of PS includes therapeutic exercise, diathermy, and local steroid injection. Among them, as radiology techniques advance, ultrasound-guided piriformis injection becomes popular for diagnosis block and treatment. Nowadays, extracorporeal shockwave therapy has widely applied in musculoskeletal disease such as plantar fasciitis, tennis elbow, and calcific tendinitis of the shoulder. However, to the investigators best knowledge, there is no study comparing the therapeutic effect between local steroid injection and shockwave. In this study, the investigators aim to compare the effect of extracorporeal shockwave therapy with ultrasound-guided piriformis corticosteroid injection.

This is a randomized controlled trial. 70 participants will be randomly divided into shockwave group and injection group. The participant in the shockwave group will receive one time extracorporeal shockwave therapy, and injection group will receive one time ultrasound-guided piriformis muscle corticosteroid injection. After the intervention, participant in both groups will receive home-based stretch exercise. Evaluation will be performed at baseline, 1 week, and 5 weeks after intervention. Outcome measures include the pain visual analog scale (VAS), hip range of motion, change of pressure pain threshold, and Oswestry Disability Index (ODI).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20 to 80
2. Unilateral buttock involvement without leg pain or paresthesia
3. Duration of symptoms ≥1 month
4. Positive trigger point or taut band at piriformis muscle, confirmed by palpation and ultrasound examination
5. Positive FAIR (flexion, adduction, internal rotation) test
6. Positive piriformis resistive test (patient actively abducts and/or externally rotates the hip while the examiner resists these movements

Exclusion Criteria:

1. Having received hip, pelvis, or lumbar spine surgery
2. Low back pain or buttock pain due to lumbosacral spine, hip or pelvis lesion other than piriformis syndrome
3. Having received shock wave therapy or corticosteroid injection for buttock pain within the past one month
4. Neurologic deficit in in the lower limbs
5. History of drug allergy to local anesthetics or corticosteroids
6. Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The pain visual analog scale (VAS) | change between baseline and at 1 week, 5 weeks after the beginning of the treatment.
  It measures severity of pain. It is performed with a 100-mm horizontal line. The end of the left side is defined as no pain, and the end of the right side as the worst pain. Participants are requested to report the severity of buttock pain in recent one week.
Oswestry Disability Index (ODI) | change between baseline and at 1 week, 5 weeks after the beginning of the treatment.
  ODI score is used for disability evaluation. It is a self-reported questionnaire with range 0-100. It has 10 questions with an minimal clinical important difference (MCID) of 10 points, with higher scores indicating more disability. The questions include pain intensity, sleep quality, and ability to perform personal care, work, sit, walk, lift, stand, and travel.

SECONDARY OUTCOMES:
hip range of motion | change between baseline and at 1 week, 5 weeks after the beginning of the treatment.
  Internal and external rotation of the hip on the affected side will be measured with a goniometer by the study assistant. The measurement will be performed in the supine position according the standard procedure.
change of pressure pain threshold | change between baseline and at 1 week, 5 weeks after the beginning of the treatment.
  It is defined as the amount of pressure needed to shift local sensation from pressure to pain. This is measured with a digital algometer and has been shown to have excellent intrarater reliability in the gluteal region (ICC = .90), with a minimal detectable change of 3.1 N/cm2. The digital algometer, made up of a 1-cm-wide disk, will be placed at the tender point between the ischial tuberosity and the greater trochanter while the patient is lying prone. The algometer's pressure will be increased gradually (with a speed approximately 1 N/cm2 per second) until the participant reports pain. The average value of three repeated measurements is recorded.

OTHER OUTCOMES:
Patient's self evaluation | change between baseline and at 1 week, 5 weeks after the beginning of the treatment.
  At 1-week and 5-week evaluations, patients are asked to report treatment effect by themselves as the following five grades: 5. Complete relief of symptoms; 4. Much improved, no need for further treatment; 3. Mildly improved, need further treatment; 2.No improvement; 1. Worse.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu YS, Shih KS, Lin YT, Hsieh LF, Liu YF, Chen YR. Efficacy of ultrasound-guided piriformis muscle corticosteroid injection versus extracorporeal shockwave therapy in patients with piriformis syndrome: A randomized controlled trial. J Formos Med Assoc. 2025 Feb 27:S0929-6646(25)00036-1. doi: 10.1016/j.jfma.2025.01.020. Online ahead of print. PMID 40016058